CLINICAL TRIAL: NCT05750719
Title: Impact of BRCA Mutation Status on Outcome and Response to Neoadjuvant Chemotherapy (NACT) in Triple-negative Breast Cancer (TNBC) Patients.
Brief Title: BRCA and NACT in TNBC Patients
Acronym: Light-Bright
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5111
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Triple-Negative Breast Cancer
Keywords: BRCA1/2; Neoadjuvant chemotherapy; Platinum agents; Triple-Negative Breast Ccancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with early triple negative breast cancer who received neoadjuvant chemotherapy.
  Interventions: Genetic: BRCA1/2 genetic testing

INTERVENTIONS:
Genetic: BRCA1/2 genetic testing — All patients will undergo genetic testing for BRCA 1 and BRCA 2 germline mutations, employing next generation sequencing (NGS) techniques.

SUMMARY:
The goal of this observational study is to evaluate data from patients with triple-negative breast cancer (TNBC) treated with neoadjuvant chemotherapy (NACT) in order to better define the impact of germline BRCA1/2 (gBRCA1/2) mutation status on outcomes in this patient population.

The aims of the study are:

* To evaluate the rate of pathologic complete response (pCR) in patients with locally advanced TNBC who performed NACT, in relation to the mutational status of gBRCA.
* To evaluate Evaluate Event Free survival (EFS) and Overall Survival (OS) in this patients population.

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) is characterized by earlier recurrence and shorter survival compared with other types of breast cancer. Moreover, approximately 15 to 25% of all TNBC patients harbor germline BRCA (gBRCA) 1/2 mutations, which confer a more aggressive phenotype. However, TNBC seems to be particularly sensitive to chemotherapy, the so-called 'triple negative paradox'. Therefore, Neoadjuvant chemotherapy (NACT) is currently considered the preferred approach for early-stage TNBC. BRCA status has also been studied as a predictive biomarker of response to platinum compounds. Although several randomized trials investigated the addition of carboplatin to standard NACT in early-stage TNBC, the role of BRCA status remains unclear. In this retrospective analysis, data from 136 consecutive patients with Stage I-III TNBC who received standard NACT, with or without the addition of carboplatin, will be evaluated in order to define clinical features and outcomes in BRCA 1/2 mutation carriers and non-carrier controls.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age older than 18 years.
* Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy.
* Tumor lesion in the breast with a palpable size of ≥ 2 cm and/or ≥ 1.5 cm by ultrasound or magnetic resonance imaging (MRI). In case of inflammatory carcinoma, the extent of inflammation can be used as measurable lesion.
* American Joint Commission on Cancer stage II or III invasive breast cancer.
* Known estrogen (ER)- and progesterone (PgR)-receptor negative tumors.
* Known HER-2/neu negative tumors, defined as IHC 1+/2+ or SISH not amplified.
* Patients suitable for neoadjuvant chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2 or Karnowsky performance status index at least 80%.
* Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 1 month prior to registration.
* Laboratory requirements:

  * Hematology: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, Hemoglobin ≥ 10 g/dL.
  * Hepatic function: Total bilirubin < 1 x UNL, ASAT (SGOT) and ALAT (SGPT)≤ 2.5 x UNL, Alkaline phosphatase ≤ 5 UNL. Patients with ASAT and / or ALAT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL are not eligible for the study.
  * Renal function: Creatinine ≤ 2 mg/dL, < 1,25 UNL (or the calculated creatinine clearance ≥ 60 mL/min).
* Paraffin tumor tissue block made available.
* Availability to provide the set up of the histological preparations for molecular analysis.
* Negative pregnancy test (urine or serum).
* Patients must be available and compliant for treatment and follow-up.

Exclusion Criteria:

* Patients candidate for adjuvant chemotherapy.
* Evidence of distant metastasis.
* Prior chemotherapy for any malignancy.
* Prior radiation therapy for breast cancer.
* Pregnant or lactating patients.
* Inadequate general condition.
* Previous malignant disease.
* Known or suspected congestive heart failure (>NYHA I) and/or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, un- or poorly controlled arterial hypertension, rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
* History of significant neurological or psychiatric disorders that would prohibit the understanding and giving of informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with early triple negative breast cancer, suitable for neoadjuvant chemotherapy achieving and not achieving pCR.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
pathologic complete response (pCR) rate | 1 month
  pCR rate of TNBC patients receiving NACT according to germline BRCA mutational status.

SECONDARY OUTCOMES:
Event Free Survival (EFS) | 1 month
  EFS of TNBC patients receiving NACT according to germline BRCA mutational status.
Overall Survival (OS) | 1 month
  OS of TNBC patients receiving NACT according to germline BRCA mutational status.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pavese F, Capoluongo ED, Muratore M, Minucci A, Santonocito C, Fuso P, Concolino P, Di Stasio E, Carbognin L, Tiberi G, Garganese G, Corrado G, Di Leone A, Generali D, Fragomeni SM, D'Angelo T, Franceschini G, Masetti R, Fabi A, Mule A, Santoro A, Belli P, Tortora G, Scambia G, Paris I. BRCA Mutation Status in Triple-Negative Breast Cancer Patients Treated with Neoadjuvant Chemotherapy: A Pivotal Role for Treatment Decision-Making. Cancers (Basel). 2022 Sep 21;14(19):4571. doi: 10.3390/cancers14194571. PMID 36230495